CLINICAL TRIAL: NCT02499159
Title: A Randomized Controlled Trial of the Effectiveness of Liposomal Bupivacaine (Exparel) When Compared to Local Injection of Bupivacaine After Thoracoscopy
Brief Title: Pain Management in Response to Exparel vs. Standard Bupivicaine
Acronym: VATS Exparel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Mednax National Medical Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-1656
Record Dates: First submitted 2015-07-08; First posted 2015-07-16 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: Exparel; Thoracoscopy; Bupivicaine; Liposomal
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel (Experimental): Liposomal Bupivicaine (Exparel) - 266 mg, 20 mL total, diluted at surgeon's discretion, Two doses of 10 mL each, into two separate incisions, delivered via 22 gauge needle.
  Interventions: Drug: Liposomal Bupivicaine
- 0.25% standard bupivicaine (Active Comparator): Bupivicaine - 0.25%, 20 mL total. Two doses of 10 mL each, into two separate incisions, delivered via 22 gauge needle.
  Interventions: Drug: 0.25% standard bupivicaine

INTERVENTIONS:
Drug: Liposomal Bupivicaine — 266 mg, 20 mL total, diluted at surgeon's discretion, delivered by 22 gauge needle.
  Other Names: Exparel
  Arms: Exparel
Drug: 0.25% standard bupivicaine — standard 0.25% bupivacaine, 20 mL total, delivered by 22 gauge needle.
  Other Names: Bupivicaine
  Arms: 0.25% standard bupivicaine

SUMMARY:
This study is looking to evaluate the efficacy of liposomal bupivicaine (Exparel) on decreasing the amount of consumed pain medications.

Patients will be randomly selected to received either Exparel or standard bupivicaine injection during surgery. Patients will be followed up to assess pain levels using a visual pain scale, and to assess how much pain medication was consumed.

DETAILED DESCRIPTION:
Exparel is a formulation of liposomal bupivacaine that is reported to allow local anesthesia for up to 72 hours post injection.

It is the investigators' aim to follow their prior study with a randomized trial to compare local infiltration of liposomal bupivacaine at the conclusion of each procedure with injections of standard .25% bupivacaine.

Patients in group A will receive, at the end of the surgical procedure, injections of liposomal bupivacaine (Exparel) (266 mg, 20 mL, diluted at surgeon's discretion) into the thoracoscopic port incision sites and around the intercostal nerves serving that space.

Patients in group B will receive, at the end of the surgical procedure, injections of standard .25% bupivacaine into the thoracoscopic port incision sites and around the intercostal nerves serving that space.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age
* Isolated thoracoscopic procedure for therapeutic or diagnostic purposes

Exclusion Criteria:

* Previous ipsilateral thoracic surgery
* Need for operative pleurectomy or pleurodesis
* Chronic use of pain medication -narcotics or nonsteroidal antiinflammatory drugs (NSAIDs), sedatives, or hypnotics
* Allergies to bupivacaine or other local anesthetics, narcotics, NSAIDs or acetaminophen
* Liver dysfunction (INR > 1.5, albumin < 2.8g/dl, bilirubin > 2mg/dl)
* Renal dysfunction (eGFR < 60ml/min/1.73m2)
* History of peptic ulcerative disease
* Severe chronic obstructive pulmonary disease (COPD) requiring continuous oxygen supplementation
* Inability to consent
* Pregnancy
* Need for conversion from a Video-Assisted Thoracic Surgery procedure to a thoracotomy
* Patient is discharged from the hospital with a chest tube in place
* Patient fails to comply with post-operative instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep J Khandhar, MD, Principal Investigator — Cardiac, Vascular, and Thoracic Surgery Associates
Locations (2):
- United States (2):
  - Cardiac, Vascular, and Thoracic Surgery Associates, Falls Church, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Background] Whitson BA, Groth SS, Duval SJ, Swanson SJ, Maddaus MA. Surgery for early-stage non-small cell lung cancer: a systematic review of the video-assisted thoracoscopic surgery versus thoracotomy approaches to lobectomy. Ann Thorac Surg. 2008 Dec;86(6):2008-16; discussion 2016-8. doi: 10.1016/j.athoracsur.2008.07.009. PMID 19022040
- [Background] Allen MS, Halgren L, Nichols FC 3rd, Cassivi SD, Harmsen WS, Wigle DA, Shen KR, Deschamps C. A randomized controlled trial of bupivacaine through intracostal catheters for pain management after thoracotomy. Ann Thorac Surg. 2009 Sep;88(3):903-10. doi: 10.1016/j.athoracsur.2009.04.139. PMID 19699918
- [Background] Chan VW, Chung F, Cheng DC, Seyone C, Chung A, Kirby TJ. Analgesic and pulmonary effects of continuous intercostal nerve block following thoracotomy. Can J Anaesth. 1991 Sep;38(6):733-9. doi: 10.1007/BF03008451. PMID 1914056
- [Background] Debreceni G, Molnar Z, Szelig L, Molnar TF. Continuous epidural or intercostal analgesia following thoracotomy: a prospective randomized double-blind clinical trial. Acta Anaesthesiol Scand. 2003 Oct;47(9):1091-5. doi: 10.1034/j.1399-6576.2003.00208.x. PMID 12969101
- [Background] Kaiser AM, Zollinger A, De Lorenzi D, Largiader F, Weder W. Prospective, randomized comparison of extrapleural versus epidural analgesia for postthoracotomy pain. Ann Thorac Surg. 1998 Aug;66(2):367-72. doi: 10.1016/s0003-4975(98)00448-2. PMID 9725371
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2004 Jun;100(6):1573-81. doi: 10.1097/00000542-200406000-00033. No abstract available. PMID 15166580

RESULTS

PARTICIPANT FLOW:
Period: Randomization
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Started | 50 | 50
Completed | 49 | 49
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: 30-Day Follow-Up Phone Call
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Started | 49 | 49
Completed | 42 | 47
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal due to ineligibility | 2 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two patients who were enrolled were not randomized due to screen failing after consent. These two patients are not included in the baseline population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | 0.25% Standard Bupivicaine | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10.9) | 65 (10.8) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 21 | 22 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 36 | 41 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Overall Amounts of Pain Medications Consumed Through Post-operative Day 7
Description: Using questionnaires, patients are asked if they took Dilaudid, Tylenol, Motrin, or other opioids and if so, how many tablets.
Time Frame: Assessed daily for 7 days post-procedure
Population: 4 participants from the Exparel group and 6 participants from the standard group did not return a questionnaire.
Measure: Number; unit: tablets
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 45 | 44
tablets | 1294 | 1455.5

2. Secondary Outcome: Scores on a Analog Pain Scale (7 Days)
Description: Using questionnaires, patients are asked what their pain level is based on a scale from 0-10, 10 being the absolute worst pain and 0 being no pain.
Time Frame: Assessed at day 7 post-procedure
Measure: Median (Inter-Quartile Range); unit: Median score on postoperative day 7
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 49 | 49
Median score on postoperative day 7 | 1.5 [1 to 3] | 1 [0 to 2]

3. Secondary Outcome: Scores on an Analog Pain Scale (30 Days)
Description: as for outcome 2
Time Frame: Assessed at 30 days post-procedure
Population: 42 subjects in the Exparel group and 47 subjects in the standard group completed the 30-day survey.
Measure: Median (Inter-Quartile Range); unit: Median score on postoperative day 30
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 42 | 47
Median score on postoperative day 30 | 0 [0 to 0] | 0 [0 to 0.5]

4. Secondary Outcome: Number of Patients With Paresthesias (Postoperatively at 7 Days)
Description: Patients are asked if they have experienced a pricking or tingling sensation caused by potential pressure or damage to peripheral nerves since the procedure.
Time Frame: Assessed at day 7 post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 49 | 49
Participants | 10 | 20

5. Secondary Outcome: Proportion of Patients With Paresthesias (Postoperatively at 30 Days)
Description: Patients are asked if they have experienced a pricking or tingling sensation caused by potential pressure or damage to peripheral nerves
Time Frame: Assessed at day 30 post-procedure
Population: 42 subjects in the Exparel group and 47 subjects in the standard group completed the 30-day survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 42 | 47
Participants | 6 | 5

6. Secondary Outcome: Hospital Length of Stay
Description: Median length of stay in days until discharge.
Time Frame: From end of procedure until discharge, usually 0-2 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 49 | 49
days | 0 [0 to 1] | 0 [0 to 1]

7. Secondary Outcome: Return to Baseline Activity
Description: Using surveys, patients are asked if they have been able to return to baseline activity levels.
Time Frame: Assessed at 30 days post-procedure
Population: 42 subjects in the Exparel group and 47 subjects in the standard group completed the 30 day survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 42 | 47
Participants | 40 | 47

8. Secondary Outcome: Return to Work
Description: Using surveys, patients are asked if they have been able to return to work.
Time Frame: Assessed at 30 days post-procedure
Population: 42 subjects in the Exparel group and 47 patients in the standard group completed the 30-day survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 42 | 47
Participants | 24 | 17

9. Secondary Outcome: Days Until Return to Work
Description: Using surveys, the number of days to return to work was assessed for patients who were able to return to work.
Time Frame: Assessed at 30 days post-procedure
Population: At the 30-day call, 24 subjects in the Exparel group and 17 subjects in the standard group indicated that they were able to return to work. Number of days were assessed for these subjects.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 24 | 17
days | 6.5 [3 to 10] | 5 [4 to 7]

10. Secondary Outcome: Overall Hospital Cost
Description: Overall hospital cost of patient procedure and stay will be assessed.
Time Frame: Total cost assessed from patient registration until discharge to home (usually 0-2 days).
Population: Data on hospital cost was not collected.
Arm/Group | Exparel | 0.25% Standard Bupivicaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From procedure until the 30-day (plus or minus 10 days) post-procedure phone call.
Arm/Group | Exparel | 0.25% Standard Bupivicaine
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/49
Other Adverse Events (participants affected / at risk) | 5/49 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=49) | 0.25% Standard Bupivicaine (N=49)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Anxiety
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=49) | 0.25% Standard Bupivicaine (N=49)
Amaurosis Fugax (Nervous system disorders) | 1 (1) | 0 (0)
Nose bleeds (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Urinary blockage (Renal and urinary disorders) | 1 (1) | 0 (0)
Brain tumor (Nervous system disorders) | 1 (1) | 0 (0)
Occipital Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT02499159/Prot_SAP_000.pdf